CLINICAL TRIAL: NCT01566435
Title: Phase II Trial of Nab-Paclitaxel, Cisplatin, and 5-FU (ACF) as Induction Therapy Followed by Definitive Concurrent Chemoradiation for Locally Advanced Squamous Cell Carcinoma of the Head and Neck (HNSCC)
Brief Title: Induction Chemotherapy With ACF Followed by Chemoradiation Therapy for Adv. Head & Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201202113
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Results first posted 2015-12-14 (Estimated); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Taxes; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; Nanoparticles; Cisplatin; Fluorouracil; Radiotherapy, Intensity-Modulated; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1-ACF Induction Therapy Followed by Chemoradiation Therapy (Experimental): ACF Induction Therapy (Cycle 1 and Cycle 2 - each cycle is every 3 weeks)
  1. nab-Paclitaxel 100 mg/m^2 on Days 1, 8, and 15
  2. Cisplatin 75 mg/m^2 on Day 1
  3. 5-FU 750 mg/m^2 on Days 1-3
  If patient has complete or partial response, he/she will receive an additional ACF cycle (cycle 3). If patient has stable disease or progressive disease will not receive the third cycle of ACF.
  Definitive Therapy
  1. Cisplatin 100 mg/m^2 IV on Days 1, 22, and 43
  2. Intensity modulated radiation therapy (IMRT) 7000 cGy in 35 fractions of 200 cGy each over 7 weeks. A dose of 6300 cGy in 35 fractions is optional and may be delivered to area considered to be at intermediate risk. Additional regions in the ipsilateral and contralateral neck at risk for microscopic disease in the cervical lymph nodes will receive 5600 cGy in 35 fractions.
  3. If patient cannot receive cisplatin then he/she will receive cetuximab 250 mg/m^2 IV week for 8 weeks
  Interventions: Drug: paclitaxel albumin-stabilized nanoparticle formulation; Drug: Cisplatin; Drug: Fluorouracil; Radiation: Intensity modulated radiation therapy; Drug: Cetuximab; Procedure: Quality-of-life assessment

INTERVENTIONS:
Drug: paclitaxel albumin-stabilized nanoparticle formulation
  Other Names: ABI-007; Abraxane; Albumin-Stabilized Nanoparticle Paclitaxel; nab paclitaxel; nab-paclitaxel, nanoparticle
Drug: Cisplatin
  Other Names: CACP; CDDP; CPDD; DDP; Neoplatin
Drug: Fluorouracil
  Other Names: 5-fluorouracil, 5-Fluracil, 5-FU, Adrucil, Efudex, FU
Radiation: Intensity modulated radiation therapy
  Other Names: IMRT
Drug: Cetuximab
  Other Names: Anti-EGFR Monoclonal Antibody, C225, C225 monoclonal antibody, IMC-C225, MOAB C225, monoclonal antibody C225
Procedure: Quality-of-life assessment — ACF baseline, IMRT baseline, Day 7, Week 12, months 6 and 12
  Other Names: FACT H&N; FACT/GOG-NTX-4

SUMMARY:
This phase II trial studies the safety and effectiveness of an induction chemotherapy (ACF) consisting of paclitaxel albumin-stabilized nanoparticle formulation (nab-paclitaxel), cisplatin and fluorouracil followed by chemoradiation therapy in treating patients with stage III-IV squamous cell cancer of the head and neck. ACF may be an effective way to reduce or downgrade locally aggressive tumors, and improve the chance of eradication by chemoradiation.

DETAILED DESCRIPTION:
Compared to the standard induction regimen of TPF (docetaxel, cisplatin, and 5-FU), the ACCF (nab-paclitaxel, cisplatin, cetuximab, and 5-FU) regimen included two therapeutic changes: nab-paclitaxel was substituted for docetaxel and cetuximab was added. The investigators propose to eliminate cetuximab from the ACCF regimen to isolate the treatment effects of nab-paclitaxel when given with cisplatin and 5-FU. The primary objective of the ACF proposal is to determine the complete (CR) rate by clinical examination at the primary tumor site following two cycles of ACF. An important secondary objective will be to compare the tumor response rates at the primary site following two cycles of ACF to our historical experience following two cycles of ACCF (protocol # ABX 218/HRPO# 08-0911). In addition, the investigators will compare adverse events (AEs) between patients who receive ACF to the historical group given ACCF. From these two comparisons, we aim to determine if either ACF or ACCF is superior based on a balance of efficacy (using the surrogate prognostic endpoint of CR rate at primary tumor site) and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have selected stage III or IVa/b head and neck squamous cell carcinoma (HNSCC); all patients must have T2-T4 primary tumors; (patients with T1 tumors will be excluded); although most of these patients will have regional nodal disease, patients with no nodal disease will also be eligible
* Patient must have disease at the oropharynx, hypopharynx, larynx, or oral cavity sub-sites
* Patient must have measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 10 mm with CT scan
* Patient must be >= 18 years of age.
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Patient must have adequate bone marrow and organ function as defined below:

  * Absolute neutrophil count (ANC) >= 1500/mcL
  * Platelets > 100,000/mcL
  * Hemoglobin > 9.0 g/dL
  * Total bilirubin =< 1.5 mg/dL
  * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN)
  * Alkaline phosphatase =< 2.5 x ULN
  * Serum creatinine < 1.8 mg/dL
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry, for the duration of study participation, and for 3 months after completing treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately
* Patient must be able to understand and willing to sign an Institutional Review Board (IRB)-approved written informed consent document
* Patient with uncontrolled diabetes or fasting blood glucose level of greater than 200 mg/dL will be eligible for enrollment but will not be evaluable for PET imaging

Exclusion Criteria:

* Patient must not have had prior chemotherapy, prior epidermal growth factor receptor (EGFR) targeted therapy, or prior radiation therapy for HNSCC
* Patient must not have disease at the nasopharyngeal, sinus, or other sub-site not specified in the inclusion criteria; patient must not have unknown primary squamous cell carcinoma of the head and neck
* Patient must not have a history of prior invasive malignancy diagnosed within 3 years prior to study enrollment other than local stage non-melanoma skin cancer
* Patient must not be receiving any other investigational agents
* Patient must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to any of the agents used in this study
* Patient must not be taking cimetidine or allopurinol. If currently taking either of these medications, patient must discontinue for one week before receiving treatment with nab-paclitaxel
* Patient must not have an uncontrolled intercurrent illness including, but not limited to, ongoing or active serious infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or serious psychiatric illness/social situations that would limit compliance with study requirements
* Patient must not be pregnant and/or breastfeeding; a negative serum or urine pregnancy test is required at screening for all female patients of childbearing potential
* Patient must not be known to be human immunodeficiency virus (HIV)-positive on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with the study agents; in addition, these patients are at increased risk of lethal infections when treated with marrow suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Patient must not have peripheral neuropathy > grade 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-08-09 (Actual); Primary Completion 2013-10-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Adkins, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adkins D, Ley J, Oppelt P, Gay HA, Daly M, Paniello RC, Jackson R, Pipkorn P, Rich J, Zevallos J, Trinkaus K, Thorstad W. Impact on Health-Related Quality of Life of Induction Chemotherapy Compared With Concurrent Cisplatin and Radiation Therapy in Patients With Head and Neck Cancer. Clin Oncol (R Coll Radiol). 2019 Sep;31(9):e123-e131. doi: 10.1016/j.clon.2019.05.007. Epub 2019 May 28. PMID 31147146
- [Derived] Adkins D, Ley J, Oppelt P, Wildes TM, Gay HA, Daly M, Rich J, Paniello RC, Jackson R, Pipkorn P, Nussenbaum B, Trinkaus K, Thorstad W. nab-Paclitaxel-based induction chemotherapy with or without cetuximab for locally advanced head and neck squamous cell carcinoma. Oral Oncol. 2017 Sep;72:26-31. doi: 10.1016/j.oraloncology.2017.07.001. Epub 2017 Jul 8. PMID 28797458
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 08/09/2012 and closed to participant enrollment on 11/07/2013.
Groups:
- Arm 1-ACF Induction Therapy Followed by Chemoradiation Therapy: ACF Induction Therapy (Cycle 1 and Cycle 2 - each cycle is every 3 weeks)
  * nab-Paclitaxel 100 mg/m^2 on Days 1, 8, and 15
  * Cisplatin 75 mg/m^2 on Day 1
  * 5-FU 750 mg/m^2 on Days 1-3
  If patient has complete or partial response, he/she will receive an additional ACF cycle (cycle 3). If patient has stable disease or progressive disease will not receive the third cycle of ACF.
  Definitive Therapy
  * Cisplatin 100 mg/m^2 IV on Days 1, 22, and 43
  * Intensity modulated radiation therapy (IMRT) 7000 cGy in 35 fractions of 200 cGy each over 7 weeks. A dose of 6300 cGy in 35 fractions is optional and may be delivered to area considered to be at intermediate risk. Additional regions in the ipsilateral and contralateral neck at risk for microscopic disease in the cervical lymph nodes will receive 5600 cGy in 35 fractions.
  * If patient cannot receive cisplatin then he/she will receive cetuximab 250 mg/m^2 IV week for 8 weeks
Period: ACF Induction Therapy
Arm/Group | Arm 1-ACF Induction Therapy Followed by Chemoradiation Therapy
Started | 30
Completed | 30
Not Completed | 0
Period: ACF Definitive Chemoradiation-cisplatin
Arm/Group | Arm 1-ACF Induction Therapy Followed by Chemoradiation Therapy
Started | 28
Completed | 27
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: ACF Definitive Chemoradiation-cetuximab
Arm/Group | Arm 1-ACF Induction Therapy Followed by Chemoradiation Therapy
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1-ACF Induction Therapy Followed by Chemoradiation Therapy: ACF Induction Therapy (Cycle 1 and Cycle 2 - each cycle is every 3 weeks)
  1. nab-Paclitaxel 100 mg/m2 on Days 1, 8, and 15
  2. Cisplatin 75 mg/m2 on Day 1
  3. 5-FU 750 mg/m2 on Days 1-3
  If patient has complete or partial response, he/she will receive an additional ACF cycle (cycle 3). If patient has stable disease or progressive disease will not receive the third cycle of ACF.
  Definitive Therapy
  1. Cisplatin 100 mg/m2 IV on Days 1, 22, and 43
  2. Intensity modulated radiation therapy (IMRT) 7000 cGy in 35 fractions of 200 cGy each over 7 weeks. A dose of 6300 cGy in 35 fractions is optional and may be delivered to area considered to be at intermediate risk. Additional regions in the ipsilateral and contralateral neck at risk for microscopic disease in the cervical lymph nodes will receive 5600 cGy in 35 fractions.
  3. If patient cannot receive cisplatin then he/she will receive cetuximab 250 mg/m2 IV week for 8 weeks
Arm/Group | Arm 1-ACF Induction Therapy Followed by Chemoradiation Therapy
Number analyzed (Participants) | 30
Age, Continuous [Mean (Full Range); unit: years] | 58.8 [43 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 30
Smoking history [Number; unit: participants]
  Yes | 23
  No | 7
T Stage [Number; unit: participants] — -T Stage (primary tumor)
  * T2 = Tumor > 2 cm but not more than 4 cm in greatest dimension
  * T3 = Tumor > 4 cm in greatest dimension
  * T4a = Lip - Tumor invades through cortical bone, inferior alveolar nerve, floor of mouth, or skin of face, Oral cavity - Tumor invades adjacent structures (eg, through cortical bone into deep extrinsic muscle of the tongue, maxillary sinus, or skin of face
  * T4b - Tumor invades masticator space, pterygoid plates, or skull base and/or encases internal carotid artery
  participants
    T2 | 8
    T3 | 13
    T4 | 9
Primary tumor site [Number; unit: participants]
  Oropharynx | 18
  Larynx | 9
  Hypopharynx | 3
HPV Status [Number; unit: participants]
  HPV-related OPSCC | 17
  HPV-unrelated HNSCC | 13
Overall stage of disease [Number; unit: participants] — * The pathological staging system used for oral cavity or oropharyngeal cancers is the American Joint Committee on Cancer (AJCC) TNM system.
  * Stage III is considered a better outcome than Stage IVB
  participants
    III | 3
    IVA | 18
    IVB | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response (CR) by Clinical Exam at Primary Tumor Site
Description: * Response will be assessed by laryngoscopy.
  * CR: disappearance of all lesions
Time Frame: 6 weeks (2 cycles of therapy)
Measure: Number; unit: percentage of participants
Groups:
- Arm 1 (ACF): ACF Induction Therapy (Cycle 1 and Cycle 2 - each cycle is every 3 weeks)
  1. nab-Paclitaxel 100 mg/m2 on Days 1, 8, and 15
  2. Cisplatin 75 mg/m2 on Day 1
  3. 5-FU 750 mg/m2 on Days 1-3
  If patient has complete or partial response, he/she will receive an additional ACF cycle (cycle 3). If patient has stable disease or progressive disease will not receive the third cycle of ACF.
  Definitive Therapy
  1. Cisplatin 100 mg/m2 IV on Days 1, 22, and 43
  2. Intensity modulated radiation therapy (IMRT) 7000 cGy in 35 fractions of 200 cGy each over 7 weeks. A dose of 6300 cGy in 35 fractions is optional and may be delivered to area considered to be at intermediate risk. Additional regions in the ipsilateral and contralateral neck at risk for microscopic disease in the cervical lymph nodes will receive 5600 cGy in 35 fractions.
  3. If patient cannot receive cisplatin then he/she will receive cetuximab 250 mg/m2 IV week for 8 weeks
Arm/Group | Arm 1 (ACF)
Number analyzed (Participants) | 30
percentage of participants | 76.7

2. Secondary Outcome: Percentage of Participants With Partial Response (PR) at Primary Tumor Site
Description: * Response will be assessed by laryngoscopy.
  * PR: at least 30% decrease in the sum of the longest diameter of target lesions taking as reference the baseline sum longest diameter
Time Frame: 6 weeks (2 cycles of therapy)
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 (ACF)
Number analyzed (Participants) | 30
percentage of participants | 16.7

3. Secondary Outcome: Number of Participants Per Anatomic Tumor Response by CT Scan
Description: * Response assessed using RECIST criteria version 1.0
  * Complete response: disappearance of all target lesions
  * Partial response: at least 30% decrease in the sum of the longest diameter of target lesions taking as reference the baseline sum longest diameter
  * Non-complete response/non-progression: persistence of one or more non-target lesion and/or maintenance of tumor marker level above the upper limits of normal.
  * Progression: at least a 20% increase in the sum of the LD of target lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 6 weeks (2 cycles of therapy)
Measure: Number; unit: participants
Arm/Group | Arm 1 (ACF)
Number analyzed (Participants) | 30
participants
  Complete response | 23
  Partial response | 5
  Non-complete response/Non-progression/Progression | 2

4. Secondary Outcome: Metabolic Tumor Responses as Measured by FDG-PET/CT
Description: * Complete metabolic response (CMR): Complete resolution of all metabolically active target and non-target lesions, and no interval development of new lesions
  * Partial metabolic response (PMR): 20% or greater decrease in max SUV from baseline, no metabolic progression of non-target lesions and no new lesions and/or decrease in total number of non-target lesions, no new lesions
  * Stable metabolic disease (SMD) - does not qualify for CMR, PMR, or PMD
  * Progressive metabolic disease (PMD): development of one or more metabolically active lesions or 20% or greater increased in max SUV from baseline, new metabolically active lesions
Time Frame: 6 weeks (2 cycles of therapy)
Population: 29 participants out of 30 participants were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Arm 1-ACF Induction Therapy Followed by Chemoradiation Therapy
Number analyzed (Participants) | 29
participants
  Complete metabolic response | 3
  Partial metabolic response rate | 25
  Stable or Progressive Metabolic Disease | 1

5. Secondary Outcome: Overall Survival Rate
Description: -Overall survival rate is the percentage of participants who are alive at 2 years.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 (ACF)
Number analyzed (Participants) | 30
percentage of participants | 93.0

6. Secondary Outcome: Adverse Events as Measured by Number of Participants That Experienced Each Common Adverse Event During ACF Induction Therapy
Description: Assessed by NCI-CTCAE version 3
Time Frame: From start of treatment through 30 days after end of treatment
Measure: Number; unit: participants
Arm/Group | Arm 1-ACF Induction Therapy Followed by Chemoradiation Therapy
Number analyzed (Participants) | 30
participants
  Grades 1/2 Neutropenia | 9
  Grades 3/4 Neutropenia | 7
  Grades 1/2 Thrombocytopenia | 11
  Grades1/2 Anemia | 24
  Grades 3/4 Anemia | 2
  Grades 1/2 Tinnitus | 3
  Grades 3/4 Tinnitus | 1
  Grades 1/2 Rash | 5
  Grades 1/2 Diarrhea | 9
  Grades 3/4 Diarrhea | 3
  Grades 1/2 Mucositis | 8
  Grades 3/4 Mucositis | 1
  Grades 3/4 Febrile Neutropenia | 4
  Grades 1/2 Edema: Limb | 5
  Grades 1/2 Creatinine | 7
  Grades 1/2 ALT | 4
  Grades 3/4 ALT | 1
  Grades 1/2 AST | 2
  Grades 3/4 AST | 1
  Grades 1/2 Sensory Neuropathy-peripheral | 4
  Grades 3/4 Sensory Neuropathy - peripheral | 1
  Grades 1/2 Fatigue | 13
  Grades 3/4 Fatigue | 1
  Grades 1/2 Weight Loss | 7
  Grades 3/4 Weight Loss | 6

7. Secondary Outcome: Changes in Secreted Protein Acidic and Rich in Cysteine (SPARC) Expression by Immunohistochemistry (IHC) in Primary Tumor Tissue
Description: SPARC and Ki-67 expression will be assessed at this institution by IHC stains performed on clinically available tumor specimens (paraffin blocks). The specimens will be collected retrospectively from prior biopsies (pre treatment and following 2 cycles of ACF) that will have consisted of a minimum of two needle cores (16-18 gauge) or two small incisional/excisional pieces of tumor. These will have been placed in 2% buffered formalin and transported to the surgical pathology processing lab.
Time Frame: 6 weeks (2 cycles of therapy)
Population: The data was not collected for this outcome measure.
Arm/Group | Arm 1-ACF Induction Therapy Followed by Chemoradiation Therapy
Number analyzed (Participants) | 0

8. Secondary Outcome: Complete Response (CR) or Partial Response (PR) at Regional (Neck) Nodes as Measured by Clinical Exam
Time Frame: 6 weeks (2 cycles of therapy)
Population: 2 participants were not evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Arm 1-ACF Induction Therapy Followed by Chemoradiation Therapy
Number analyzed (Participants) | 28
participants
  Complete response | 19
  Partial response | 7

9. Secondary Outcome: Changes in Ki-67 Expression by Immunohistochemistry (IHC) in Primary Tumor Tissue
Description: Ki-67 expression will be assessed at this institution by IHC stains performed on clinically available tumor specimens (paraffin blocks). The specimens will be collected retrospectively from prior biopsies (pre treatment and following 2 cycles of ACF) that will have consisted of a minimum of two needle cores (16-18 gauge) or two small incisional/excisional pieces of tumor. These will have been placed in 2% buffered formalin and transported to the surgical pathology processing lab.
Time Frame: 6 weeks (2 cycles of therapy)
Population: The data was not collected for this outcome measure.
Arm/Group | Arm 1-ACF Induction Therapy Followed by Chemoradiation Therapy
Number analyzed (Participants) | 0

10. Secondary Outcome: Disease-free Survival (DFS) Rate
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 (ACF)
Number analyzed (Participants) | 30
percentage of participants | 97.0

11. Secondary Outcome: Progression-free Survival (PFS)
Description: -Progression: at least a 20% increase in the sum of the longest diameter (LD) of target lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1-ACF Induction Therapy Followed by Chemoradiation Therapy
Number analyzed (Participants) | 30
percentage of participants | 97

12. Secondary Outcome: Quality of Life (QOL) as Measured by Functional Assessment of Cancer Therapy - Head and Neck (FACT-H&N) Total Score
Description: * Includes 39 questions: 7 in physical well-being, 6 in emotional well-being, 7 in functional well-being, and 12 in head & neck
  * Scored from 0 (not at all) to 4 (very much)
  * Higher scores indicated worse physical and emotional well-being and better social/family and functional well-being
  * The FACT-H&N Total Score (range 0-148) measures the sum of the physical, social, emotional, functional, and HNCS domains
  * The maximum score of 148 reflects the best quality of life.
Time Frame: Through one year after completion of treatment
Population: Questionnaires were not collected at some time points due to various reasons including patient decision, death, lost to follow-up, and missed by staff.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm 1-ACF Induction Therapy Followed by Chemoradiation Therapy
Number analyzed (Participants) | 30
score on a scale
  Baseline | 109.7 [99.6 to 119.8]
  End of induction: number analyzed (Participants) | 28
  End of induction | 105.8 [96.2 to 115.4]
  End of chemoradiation treatment: number analyzed (Participants) | 26
  End of chemoradiation treatment | 74.2 [67.1 to 81.3]
  3 months after completion of treatment: number analyzed (Participants) | 25
  3 months after completion of treatment | 98.4 [88.0 to 108.7]
  6 months after completion of treatment: number analyzed (Participants) | 27
  6 months after completion of treatment | 107.4 [95.7 to 119.2]
  12 months after completion of treatment: number analyzed (Participants) | 22
  12 months after completion of treatment | 114.6 [105.1 to 124.1]

13. Secondary Outcome: Quality of Life (QOL) as Measured by Functional Assessment of Cancer Therapy - Head and Neck (FACT-H&N) FACT-G Total Score
Description: * Includes 39 questions: 7 in physical well-being, 6 in emotional well-being, 7 in functional well-being, and 12 in head & neck
  * Scored from 0 (not at all) to 4 (very much)
  * Higher scores indicated worse physical and emotional well-being and better social/family and functional well-being
  * The FACT-G Total Score (range 0-108) measures the sum of the physical, social, emotional, and functional domains but excludes the HNCS domain
  * The maximum score of 108 reflects the best quality of life.
Time Frame: Through end of chemoradiation
Population: as for outcome 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm 1-ACF Induction Therapy Followed by Chemoradiation Therapy
Number analyzed (Participants) | 30
score on a scale
  Baseline | 83.8 [77.1 to 90.3]
  End of induction | 79.1 [72.3 to 85.7]
  End of chemoradiation treatment | 62.3 [57 to 67.5]

14. Secondary Outcome: Quality of Life (QOL) as Measured by Functional Assessment of Cancer Therapy - Head and Neck (FACT-H&N) Trial Outcome Index (TOI)
Description: * Includes 39 questions: 7 in physical well-being, 6 in emotional well-being, 7 in functional well-being, and 12 in head & neck
  * Scored from 0 (not at all) to 4 (very much)
  * Higher scores indicated worse physical and emotional well-being and better social/family and functional well-being
  * The FACT-H&N TOI (range 0-96) measures the total score for the physical, functional, and HNCS domains but excludes the emotional and social domains
  * The maximum score of 96 reflects the best quality of life.
Time Frame: Through end of chemoradiation
Population: as for outcome 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm 1-ACF Induction Therapy Followed by Chemoradiation Therapy
Number analyzed (Participants) | 30
score on a scale
  Baseline | 69.7 [62 to 77.5]
  End of induction | 62.3 [54.8 to 69.8]
  End of chemoradiation treatment | 34.2 [28.3 to 40.1]

ADVERSE EVENTS:
Description: Serious adverse events are all grade 3, 4, or 5 anticipated or unanticipated events per CTCAE Version 3.0.
Groups:
- ACF Induction Therapy: ACF Induction Therapy (Cycle 1 and Cycle 2 - each cycle is every 3 weeks)
  1. nab-Paclitaxel 100 mg/m^2 on Days 1, 8, and 15
  2. Cisplatin 75 mg/m^2 on Day 1
  3. 5-FU 750 mg/m^2 on Days 1-3
  If patient has complete or partial response, he/she will receive an additional ACF cycle (cycle 3). If patient has stable disease or progressive disease will not receive the third cycle of ACF.
- ACF Definitive Chemoradiation Therapy-cisplatin: Definitive Therapy
  1. Cisplatin 100 mg/m^2 IV on Days 1, 22, and 43
  2. Intensity modulated radiation therapy (IMRT) 7000 cGy in 35 fractions of 200 cGy each over 7 weeks. A dose of 6300 cGy in 35 fractions is optional and may be delivered to area considered to be at intermediate risk. Additional regions in the ipsilateral and contralateral neck at risk for microscopic disease in the cervical lymph nodes will receive 5600 cGy in 35 fractions.
- ACF Definitive Chemoradiation Therapy-cetuximab: Definitive Therapy
  1. Cetuximab 250 mg/m^2 IV weekly for 8 weeks
  2. Intensity modulated radiation therapy (IMRT) 7000 cGy in 35 fractions of 200 cGy each over 7 weeks. A dose of 6300 cGy in 35 fractions is optional and may be delivered to area considered to be at intermediate risk. Additional regions in the ipsilateral and contralateral neck at risk for microscopic disease in the cervical lymph nodes will receive 5600 cGy in 35 fractions.
Arm/Group | ACF Induction Therapy | ACF Definitive Chemoradiation Therapy-cisplatin | ACF Definitive Chemoradiation Therapy-cetuximab
Serious Adverse Events (participants affected / at risk) | 15/30 | 4/27 | 0/2
Other Adverse Events (participants affected / at risk) | 30/30 | 27/27 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACF Induction Therapy (N=30) | ACF Definitive Chemoradiation Therapy-cisplatin (N=27) | ACF Definitive Chemoradiation Therapy-cetuximab (N=2)
ALT (Investigations) | 1 | 1 | 0
AST (Investigations) | 1 | 1 | 0
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 0
Creatinine (Renal and urinary disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Febrile neutropenia (Infections and infestations) | 3 | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 0
Hemoglobin (Anemia) (Blood and lymphatic system disorders) | 2 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 5 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 4 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypotension (Cardiac disorders) | 1 | 0 | 0
Infection with grade 3 or 4 neutrophils (Infections and infestations) | 1 | 0 | 0
Leukopenia (Investigations) | 8 | 1 | 0
Lymphopenia (Investigations) | 4 | 0 | 0
Mucositis (Gastrointestinal disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Neutrophils (Neutropenia) (Investigations) | 6 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0
Platelets (Thrombocytopenia) (Infections and infestations) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Skin (cellulitis) (Infections and infestations) | 1 | 0 | 0
Taste alteration (Gastrointestinal disorders) | 1 | 0 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Weight loss (General disorders) | 7 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACF Induction Therapy (N=30) | ACF Definitive Chemoradiation Therapy-cisplatin (N=27) | ACF Definitive Chemoradiation Therapy-cetuximab (N=2)
ALT (Investigations) | 4 | 1 | 0
AST (Investigations) | 2 | 3 | 0
Abdomen NOS pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal distension/bloating (Gastrointestinal disorders) | 1 | 0 | 0
Alkaline phosphatase (Investigations) | 5 | 8 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 15 | 18 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 3 | 0
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Bilirubin (Metabolism and nutrition disorders) | 2 | 2 | 0
Blurred vision (Eye disorders) | 1 | 0 | 0
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Carciac ischemia/infarction (Cardiac disorders) | 0 | 1 | 0
Chest pain (Cardiac disorders) | 1 | 0 | 0
Cold sensations (Nervous system disorders) | 0 | 1 | 0
Colitis (Infections and infestations) | 1 | 1 | 0
Confusion (Nervous system disorders) | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 5 | 11 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 0
Creatinine (Renal and urinary disorders) | 7 | 20 | 0
Dehydration (Gastrointestinal disorders) | 0 | 16 | 1
Dermatitis associated with chemoradiation (Injury, poisoning and procedural complications) | 0 | 12 | 1
Diarrhea (Gastrointestinal disorders) | 9 | 4 | 0
Diverticulitis (Gastrointestinal disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 3 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 6 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 9 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Edema: head and neck (General disorders) | 2 | 8 | 0
Edema: limb (General disorders) | 5 | 6 | 0
Edema: tongue (General disorders) | 0 | 1 | 0
Eye NOS infection (Infections and infestations) | 0 | 3 | 0
Fatigue (General disorders) | 13 | 20 | 0
Febrile neutropenia (Infections and infestations) | 1 | 0 | 0
Fever (General disorders) | 1 | 3 | 0
Flushing (Vascular disorders) | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Glomerular filtration rate (Renal and urinary disorders) | 1 | 5 | 0
Gout (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 4 | 1 | 0
Hearing (without monitoring program) (Ear and labyrinth disorders) | 0 | 3 | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 3 | 0 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 0
Hemoglobin (Anemia) (Blood and lymphatic system disorders) | 24 | 27 | 2
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Hot flashes (Vascular disorders) | 1 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 10 | 13 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 5 | 4 | 0
Hypermagenesmia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 4 | 0
Hypertension (Vascular disorders) | 2 | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 15 | 18 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 15 | 18 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 4 | 14 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 14 | 14 | 1
Hyponatremia (Metabolism and nutrition disorders) | 14 | 20 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 6 | 0
Hypotension (Vascular disorders) | 4 | 4 | 1
INR (Investigations) | 0 | 3 | 0
Infection with normal ANC (Infections and infestations) | 0 | 3 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 0
Involuntary movement (Nervous system disorders) | 0 | 1 | 0
Leukocytes (WBC) (Investigations) | 17 | 26 | 2
Limb pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
Lymphopenia (Investigations) | 24 | 26 | 2
Mood alteration - anxiety (Psychiatric disorders) | 3 | 3 | 0
Mood alteration - depression (Psychiatric disorders) | 3 | 1 | 0
Motor neuropathy (Nervous system disorders) | 0 | 1 | 0
Mucositis (Gastrointestinal disorders) | 8 | 22 | 0
Muscle weakness - whole body/generalized (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
Musculoskeltal cramping (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 9 | 16 | 0
Neutrophils (Neutropenia) (Investigations) | 10 | 15 | 0
Oral candidiasis (Infections and infestations) | 3 | 4 | 0
Oral cavity hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Oral cavity pain (Gastrointestinal disorders) | 4 | 2 | 0
PTT (Investigations) | 0 | 1 | 0
Pain (general) (General disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 7 | 0
Platelets (Thrombocytopenia) (Investigations) | 11 | 20 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 8 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5 | 3 | 0
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 4 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Rigors/chills (General disorders) | 5 | 0 | 0
Salivary gland changes (Gastrointestinal disorders) | 0 | 7 | 0
Seborrheic keratotic lesions (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Sinus drainage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 3 | 3 | 0
Skin (cellulitis) (Infections and infestations) | 0 | 2 | 0
Sweating (General disorders) | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Taste alteration (Gastrointestinal disorders) | 4 | 10 | 1
Throat/pharynx/larynx pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 1 | 3 | 1
Tinnitus (Ear and labyrinth disorders) | 4 | 7 | 1
Triglycerides, high (Investigations) | 0 | 2 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Upper airway infection NOS (Infections and infestations) | 1 | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1 | 0
Urinary tract infection NOS (Infections and infestations) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 13 | 0
Weight loss (General disorders) | 6 | 22 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes